CLINICAL TRIAL: NCT05874622
Title: A Randomized, Double-blind, Dose-escalating, Placebo-controlled Phase Ib Clinical Study of VC005 Tablets in Subjects With Rheumatoid Arthritis.
Brief Title: A Phase I Clinical Study of VC005 Tablets in Subjects With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VC005-103
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- VC005 Tablets Low Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets Medium Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets High Dose groups (Experimental)
  Interventions: Drug: VC005 tablets
- VC005 Tablets Placebo Low Dose groups (Experimental)
  Interventions: Drug: VC005 Tablets Placebo
- VC005 Tablets Placebo Medium Dose groups (Experimental)
  Interventions: Drug: VC005 Tablets Placebo
- VC005 Tablets Placebo High Dose groups (Experimental)
  Interventions: Drug: VC005 Tablets Placebo

INTERVENTIONS:
Drug: VC005 tablets — VC005 groups repeat administration for 4 weeks
  Arms: VC005 Tablets High Dose groups; VC005 Tablets Low Dose groups; VC005 Tablets Medium Dose groups
Drug: VC005 Tablets Placebo — VC005 placebo groups repeat administration for 4 weeks
  Arms: VC005 Tablets Placebo High Dose groups; VC005 Tablets Placebo Low Dose groups; VC005 Tablets Placebo Medium Dose groups

SUMMARY:
This is a randomized, double-blind, dose-escalating, placebo-controlled phase Ib clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or his/her guardian understands and voluntarily signs the informed consent form (ICF);
2. The age at the time of signing the ICF is between 18 and 70 years (including borderline values), regardless of gender;
3. A body mass index [BMI = weight (kg)/height 2 (m2)] of 18 ~30 kg/m2 at the time of screening;
4. Rheumatoid arthritis diagnosed according to the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 rheumatoid arthritis (RA) classification criteria and at least 3 months of disease duration at the time of the screening visit;
5. A diagnosis of moderately or severely active RA;
6. Have not used any disease-modifying antirheumatic drugs (DMARDs) prior to the first dose of the trial, or have been on a stable dose of methotrexate (MTX) for ≥4 weeks prior to the first dose, or have used methotrexate, salbutamol, or a dose of a drug such as methotrexate. (SASP), chloroquine/hydroxychloroquine, gold, penicillamine, etc., but had stopped using them for ≥3 weeks before the first dose. have stopped using the drug for ≥ 3 months;
7. Subjects who have been stable on NSAIDs prior to the first dose must have had a fixed drug class and a stable dose for ≥4 weeks and continue at a stable dose for the duration of the clinical trial;
8. Subjects who have been stable on oral glucocorticoids prior to the first dose must have been stable for ≥4 weeks at a dose of ≤10 mg/day (prednisone or equivalent dose of other glucocorticoids) and continue at a stable dose for the duration of the clinical trial;
9. The subject is able to communicate well with the investigator and is willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. The subjects who are allergic to the study drug or any of the components of the study drug, or are allergic (multiple drug and food allergies);
2. The subjects have used any of the following medications or treatments:

   Tyrosine kinase (JAK) inhibitor class drugs, within 1 month prior to randomization/biologic disease-modifying antirheumatic drugs (bDMARDs) within 5 half-lives prior to randomization or within 3 months,etc；
3. The subjects have a history or evidence of any of the following diseases:

   Presence of any systemic inflammatory disease other than RA (except secondary dry syndrome)/lymphoproliferative disease, etc;
4. The presence of any abnormal laboratory test at screening that meets the following criteria (not allowed to receive within 2 weeks prior to screening) Any medical support therapy such as leukocyte boosting, anemia improvement, liver protection and enzyme reduction, blood transfusion, etc;
5. Positive hepatitis B surface antigen (HBsAg) or negative hepatitis B surface antigen, negative hepatitis B surface antibody, positive hepatitis B core antibody (HBcAb) with hepatitis B virus honeybee venom(HBV)-DNA test results above the lower limit of detection; positive hepatitis C antibody (HCVAb) with hepatitis C virus ribonucleic acid (HCV-RNA) test results above the lower limit of detection; positive syphilis spirochete antibody (TPAb) ，etc;
6. Screening period ECG corrected QT interval(QTC): > 470 ms for men and > 480 ms for women, or abnormalities of clinical significance that, in the judgment of the investigator, preclude enrollment;
7. Those with a history of substance abuse or drug use within the past five years;
8. Those who have a positive urine drug screen or alcohol screen;
9. Female patients who are planning to become pregnant or who are pregnant or breastfeeding, or who are unable to use effective contraception throughout the trial and for 6 months after the trial ends;
10. Who, for any reason, are deemed by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Peak time in plasma(Tmax) | Day1、Day8、Day15、Day22、Day28
Peak Plasma Concentration (Cmax） | Day1、Day8、Day15、Day22、Day28

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University; Nanya Wang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China